CLINICAL TRIAL: NCT02589431
Title: Comparison of Total, Salivary and Calculated Free Cortisol Levels in Patients With Severe Sepsis
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, ZULEYHA KARACA, Associate professor, TC Erciyes University
Other Study IDs: TST-10-2929
Record Dates: First submitted 2015-10-20; First posted 2015-10-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Severe Sepsis
Keywords: hypothalamo pituitary adrenal axis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with severe sepsis
- Controls: Healthy subjects

SUMMARY:
Background: The purpose of the present study was to compare serum total cortisol (STC), salivary cortisol (SaC) and calculated free cortisol (cFC) levels at the baseline and after the ACTH stimulation test, in patients with severe sepsis (SS) and to determine the suitability of SaC and cFC levels instead of STC for the diagnosis of adrenal insufficiency in patients with SS.

Methods: Thirty patients with SS (15 men, and 15 women) were compared with 16 healthy controls. Low dose ACTH stimulation test (1 µg) was performed on the first, 7th and 28th days of diagnosis of SS. STC and SaC levels were measured during ACTH stimulation test.

DETAILED DESCRIPTION:
More than 90% of circulating cortisol is predominantly bound to cortisol binding globulin (CBG), but also albumin. Thus, in the presence of both hypoalbuminemia and decreased CBG levels, the ratio of bound to free cortisol levels can be altered. In this situation, measurement of FC becomes more important. Direct FC measurement is time consuming and non-automated. Thus, some indirect methods to determine FC levels had been introduced. The Coolens' method may be practical to determine FC, it estimates FC levels from STC and CBG levels. In patients with CI, the synthesis of CBG and albumin is reduced leading to overestimation of adrenal insufficiency if we only use STC levels. Since some studies demonstrated that salivary cortisol (SaC) reflect free or unbound plasma cortisol levels, this method is used more often in clinical studies. STC and SaC levels at baseline and after ACTH stimulation had been used in some studies in patients with critical illness.

The aim of the present study was to compare STC, SaC and calculated free cortisol (cFC) levels at baseline and after the ACTH stimulation test in patients with SS and determine the suitability of SaC and cFC levels instead of STC for the diagnosis of adrenal insufficiency in patients with SS. And secondary aims of this study was to compare these parameters in patients with SS with healthy controls and check their effects on survival status of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe sepsis.

Exclusion Criteria:

* Diabetes Mellitus,
* Pregnancy, and
* Use of glucocorticoids of any kind.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thirthy patients with severe sepsis (15 men, and 15 women), and 16 (8 men and 8 women) healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Total Salivary and Calculated Free Cortisol Levels In Patients With Severe Sepsis | 24 months
  Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Medical School Department of Endocrinology, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Background] Cooper MS, Stewart PM. Corticosteroid insufficiency in acutely ill patients. N Engl J Med. 2003 Feb 20;348(8):727-34. doi: 10.1056/NEJMra020529. No abstract available. PMID 12594318
- [Background] Annane D, Bellissant E. Prognostic value of cortisol response in septic shock. JAMA. 2000 Jul 19;284(3):308-9. No abstract available. PMID 10891961
- [Background] Marik PE, Pastores SM, Annane D, Meduri GU, Sprung CL, Arlt W, Keh D, Briegel J, Beishuizen A, Dimopoulou I, Tsagarakis S, Singer M, Chrousos GP, Zaloga G, Bokhari F, Vogeser M; American College of Critical Care Medicine. Recommendations for the diagnosis and management of corticosteroid insufficiency in critically ill adult patients: consensus statements from an international task force by the American College of Critical Care Medicine. Crit Care Med. 2008 Jun;36(6):1937-49. doi: 10.1097/CCM.0b013e31817603ba. PMID 18496365
- [Background] Annane D, Maxime V, Ibrahim F, Alvarez JC, Abe E, Boudou P. Diagnosis of adrenal insufficiency in severe sepsis and septic shock. Am J Respir Crit Care Med. 2006 Dec 15;174(12):1319-26. doi: 10.1164/rccm.200509-1369OC. Epub 2006 Sep 14. PMID 16973979
- [Background] Dickstein G. High-dose and low-dose cosyntropin stimulation tests for diagnosis of adrenal insufficiency. Ann Intern Med. 2004 Feb 17;140(4):312-3; author reply 313-4. doi: 10.7326/0003-4819-140-4-200402170-00026. No abstract available. PMID 14970166
- [Background] Hamrahian AH, Oseni TS, Arafah BM. Measurements of serum free cortisol in critically ill patients. N Engl J Med. 2004 Apr 15;350(16):1629-38. doi: 10.1056/NEJMoa020266. PMID 15084695
- [Background] Coolens JL, Van Baelen H, Heyns W. Clinical use of unbound plasma cortisol as calculated from total cortisol and corticosteroid-binding globulin. J Steroid Biochem. 1987 Feb;26(2):197-202. doi: 10.1016/0022-4731(87)90071-9. PMID 3560936
- [Background] Deutschbein T, Unger N, Mann K, Petersenn S. Diagnosis of secondary adrenal insufficiency: unstimulated early morning cortisol in saliva and serum in comparison with the insulin tolerance test. Horm Metab Res. 2009 Nov;41(11):834-9. doi: 10.1055/s-0029-1225630. Epub 2009 Jul 7. PMID 19585406
- [Background] Gozansky WS, Lynn JS, Laudenslager ML, Kohrt WM. Salivary cortisol determined by enzyme immunoassay is preferable to serum total cortisol for assessment of dynamic hypothalamic--pituitary--adrenal axis activity. Clin Endocrinol (Oxf). 2005 Sep;63(3):336-41. doi: 10.1111/j.1365-2265.2005.02349.x. PMID 16117823
- [Derived] Elbuken G, Karaca Z, Tanriverdi F, Unluhizarci K, Sungur M, Doganay M, Kelestimur F. Comparison of total, salivary and calculated free cortisol levels in patients with severe sepsis. J Intensive Care. 2016 Jan 8;4:3. doi: 10.1186/s40560-015-0125-0. eCollection 2016. PMID 26753096